CLINICAL TRIAL: NCT06798688
Title: Software Algorithm Using Machine Learning and Threshold Based Methods for Predicting Exacerbations and Deterioration
Brief Title: In This Study, the Sponsor Would Like to Collaborate with Institution and Investigator to Aggregate Participants Data and to Pilot Its Software Algorithm Using Machine Learning and Threshold Based Methods for Predicting Exacerbations and Deterioration Within a 60 Days Period Post-discharge
Status: Not yet recruiting | Type: Observational
Sponsor: Respiree Pte Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 2025-001
Record Dates: First submitted 2025-01-22; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: A non-invasive cardio-respiratory sensor will be applied on the subjects to measure parameters to identify exacerbations — This Study aims to pilot software algorithms based on respiratory features and hemodynamics for predicting exacerbations on a total of 20 participants with COPD. The end-points of this Study includes the following:
  1. To validate respiratory-based biomarkers in models to predict exacerbations - benchmarking to be done versus physician assess exacerbations, emergency department visits, hospitalizations and any other visit.
  2. To validate level of compliance, drop-out rate and if additional measures are required to get participants to follow-on

SUMMARY:
In this study, the sponsor would like to collaborate with Institution and Investigator to aggregate participants data and to pilot its software algorithm using machine learning and threshold based methods for predicting exacerbations and deterioration within a 60 days period post-discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age 18 or older
2. Receives all primary and specialty care at Institution
3. Participants will be enrolled at discharge (and not designate hospital or ED)
4. A history of one of the following diagnoses:

   a. c. Chronic obstructive pulmonary disease
5. At least two documented exacerbations of the above disease in the past 12 months as defined by the following corresponding criteria:

   a. Chronic obstructive pulmonary disease exacerbation: all three of (1) increase in frequency and severity or severity of cough, (2) increase in volume and/or change of character of sputum production, and (3) increase in dyspnea, and requiring treatment with short-acting bronchodilators, antibiotics, and oral or intravenous glucocorticoids.
6. Participants able to provide informed consent.
7. Participants will be enrolled at discharge (and not designate hospital or ED)

Exclusion Criteria:

1. Participants with neuromuscular diseases and seizures
2. Participants enrolled in hospice care or life expectancy less than three months.
3. Participants living more than 60 miles away from Institution and Investigator
4. Participants with expected out of state travel within a 30-day period or travel to a location with no internet access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The enrolment goal is 20 participants with at least 2 documented exacerbations in the past 12 months for a period of 8 weeks each. In addition to the baseline visit and Study on-boarding, there will be 2 follow-ups every month. Participants will be enrolled at discharge (and not designate hospital or ED).
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Identifying readmissions using respiratory biomarkers | 60-days
  To validate respiratory-based biomarkers in models to predict exacerbations - benchmarking to be done versus physician assess exacerbations, emergency department visits, hospitalizations and any other visit.

SECONDARY OUTCOMES:
Validate compliance and usability | 60-days
  To validate level of usability using self-assessed questionnaires required to get participants to follow-on

IPD SHARING:
Plan to Share IPD: No